CLINICAL TRIAL: NCT01503853
Title: Discussing Costs in the Doctor-Patient Encounter
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911133; 11-CH-N133
Record Dates: First submitted 2011-12-31; First posted 2012-01-04 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-09-16

CONDITIONS: Chronic Illness; Financial Burden
Keywords: Medical Costs; Health Care; Focus Groups
MeSH Terms: conditions — Chronic Disease; Financial Stress

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- The costs of medical care have a major effect on patients during illness and treatment. Surveys with patients and doctors show that both are interested in discussing the costs of treatment. But they rarely talk about these issues. Both worry about whether it is appropriate to discuss financial matters in the clinical setting. They are also concerned about whether this topic will be an awkward one. Researchers are interested in studying how people want their doctors to talk to them about the costs of illness and medical care.

Objectives:

- To explore and better understand patients views on whether and how doctors should talk about the costs of illness and medical care.

Eligibility:

- English- or Spanish-speaking adults (at least 18 years of age) who are covered by health insurance.

Design:

* Participants will be asked to take part in a 2 1/2-hour focus group. Ten to 12 people will come together to discuss their thoughts and opinions.
* A member of the research team will lead the group discussion. The leader will ask a list of questions about health care payment issues. Those in the focus group will discuss these issues.
* Participants will receive a small cash payment and a light snack.

DETAILED DESCRIPTION:
BACKGROUND:

The cost of illness and medical care has profound implications for society as a whole and for individual patients as they experience being sick and seeking treatment. It is both appropriate and imperative that these costs be discussed in the doctor-patient encounter. Surveys with patients and doctors show that both parties have the desire to discuss costs, yet they rarely have these conversations because of worries about the appropriateness and potential awkwardness of discussing financial matters in the clinical encounter.

In the existing literature we find that patients express a preference for more care, newer care, and expensive care (as they believe cost indicates better care), and they react negatively to conversations they perceive as encouraging rationing. Yet rationing - the use of allocation criteria to distribute resources - is inevitable when resources are limited, and acceptable when done fairly. Recognizing the need for bedside rationing and endeavoring to promote bedside rationing are not antithetical to patient-centered care, however. Open and honest conversations about rationing, when carried out appropriately, can be consistent with patient-centered care and the view of patients as moral agents.

Patients resistance to discussions of rationing, coupled with the financial burden of illness and the reality of rising health care costs, all point to the pressing need to explore strategies for how physicians can address costs in ways that are understanding, empathic, and palatable to patients. In the literature we find scant empirical evidence about how patients would react to doctors talking about (and considering) costs. This study seeks the patient perspective on how these honest conversations about costs can be carried out in a sensitive and appropriate manner.

OBJECTIVE:

This project aims to explore and better understand patients perspectives about whether and how doctors should talk about and address the costs of illness and medical care. Ultimately we hope to promote the ability of doctors to discuss and address financial issues in their encounters with patients in a way that maintains trust, advocacy and integrity.

* Participants will be more receptive to discussing personal costs than societal (pooled) costs with their physicians.
* Willingness to discuss personal cost in the clinical encounter will vary with participant socio-demographic characteristics.
* Following group discussions about addressing cost of care in the clinical encounter, participants will be more receptive to discussion of costs in the clinical encounter.
* Following group discussion, participants will be more inclined to choose less expensive care.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* RAND Corp Survey Research Group will be in charge of recruiting participants. They will work with an experienced focus group recruitment vendor to identify, screen and schedule eligible participants from the LA/Santa Monica area and the Washington DC area. Candidates for the focus groups must be individuals who are 18 years old or older, able to provide informed consent, and who speak English or Spanish well enough to participate in one of the focus groups. In addition, participants must have health insurance coverage at the time of recruitment. The focus groups will include a mix of participants in terms of gender, age, race/ethnicity, educational level, SES, and health insurance coverage type. While we will not be excluding HHS or other federal employees from participating (as we see no compelling reason to do so), we will not be recruiting predominantly HHS or other federal employees because we seek a generalizable sample.
* Participants will be either English or Spanish speaking adults. Focus groups will include participants with the following varied characteristics:
* age (working adults with and without dependents and retirees); ethnic/racial groups (African American, Latino, Non-Hispanic whites);
* varied economic status (incomes below 300% of the Federal poverty threshold, and above).
* Specifically, participants will be recruited to ensure sufficient socio-demographic representation and adequate numbers to test our study hypotheses. Because we will recruit subjects with the intention of producing generalizable results, we will not recruit disproportionate numbers of HHS or other federal employees (although these individuals will not be excluded from participation).
* After the two pilot groups, twenty focus groups each including 8-12 participants will be conducted for a maximum total of 264 participants. Of the twenty focus groups, sixteen will be conducted in English and 4 will be conducted in Spanish.
* Half of participants will have incomes under 300% of the federal poverty threshold in order to guarantee ascertainment of perspectives of participants of varied socio-economic status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2011-04-16; Study Completion 2016-09-16

CONTACTS AND LOCATIONS:
Overall Officials: Marion Danis, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- RAND, Santa Monica, California, United States

REFERENCES:
- [Background] Blendon RJ, Brodie M, Benson JM, Altman DE, Buhr T. Americans' views of health care costs, access, and quality. Milbank Q. 2006;84(4):623-57. doi: 10.1111/j.1468-0009.2006.00463.x. PMID 17096637
- [Background] Coast J. Who wants to know if their care is rationed? Views of citizens and service informants. Health Expect. 2001 Dec;4(4):243-52. doi: 10.1046/j.1369-6513.2001.00147.x. PMID 11703498
- [Background] Halpern J. What is clinical empathy? J Gen Intern Med. 2003 Aug;18(8):670-4. doi: 10.1046/j.1525-1497.2003.21017.x. PMID 12911651